CLINICAL TRIAL: NCT01136031
Title: A Phase I/II Trial of Second-line Chemotherapy With Paclitaxel and Irinotecan in Fluoropyrimidine- and Platinum-Pretreated Advanced Gastric Cancer
Brief Title: Paclitaxel and Irinotecan in Advanced Gastric Cancer
Acronym: TI-2ndAGC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0703-042-201
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Advanced Gastric Cancer
Keywords: advanced gastric cancer; 1st-line failure
MeSH Terms: interventions — Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel and irinotecan (Experimental)
  Interventions: Drug: Paclitaxel and irinotecan

INTERVENTIONS:
Drug: Paclitaxel and irinotecan — In phase I part, Level Paclitaxel (mg/m²) Irinotecan (mg/m²)
  1. 100 100
  2. 100 120
  3. 135 120
  4. 135 160
  every 3 week

SUMMARY:
* Usually the combination of fluoropyrimidine with platinum is used as a first line chemotherapy (for example, 5-FU+cisplatin, capecitabine+cisplatin, S-1+ cisplatin, 5-FU+oxaliplatin) in advanced gastric cancer.
* After failure with this combination, taxane-based regimen or irinotecan-based regimen is usually used. But, as a second-line regimen, the combination of topoisomerase inhibitor with taxane has not been fully evaluated until now.
* So we designed this phase I/II study to evaluate the efficacy and toxicity of second-line chemotherapy with paclitaxel and irinotecan in fluoropyrimidine and platinum-pretreated advanced gastric cancer.

DETAILED DESCRIPTION:
In gastric cancer, several active chemotherapeutic agents have been introduced. Fluoropyrimidine, platinum, taxane and topoisomerase inhibitor are the most commonly used agents. Many available single or combination regimens are existed. But, there is no standard palliative chemotherapy regimen as a first line treatment in unresectable advanced gastric cancer. Thereafter there is also no standard second line regimen.

Usually the combination of fluoropyrimidine with platinum is used as a first line chemotherapy (for example, 5-FU+cisplatin, capecitabine+cisplatin, S-1+ cisplatin, 5-FU+oxaliplatin). After failure with this combination, taxane-based regimen or irinotecan-based regimen is usually used. But, as a second-line regimen, the combination of topoisomerase inhibitor with taxane has not been fully evaluated until now.

In some studies using docetaxel and irinotecan combination in gastric cancer, the toxicity is highly concerned. (Jatoi A et al. 2002, Lordick F etl al. 2003, S Enrech et al. 2003, Chang HM et al. 2003) The combination of paclitaxel and irinotecan in gastric cancer is evaluated in two studies until now as far as we know (K Kobayashi et al. 2006, Hecht JR et al. 2003). These are phase I/II design and used this combination as first or second line treatment of gastric cancer. The response rate is 29.6% and 27% respectively. In one study, grade 3,4 hematologic toxicity is 33.3%. The dosing schedule is different between these two studies.

In one study, paclitaxel 50mg/m2 and irinotecan 50mg/m2 is used day 1and day 8 every 3 weeks. In the other study, paclitaxel 100mg/m2 and irinotecan 225mg/m2 is used every 3 weeks.

In these studies, the state of UGT1A1 polymorphism of enrolled patients has not been reported. Recently it is well known that the UGT1A1 polymorphism influences on the toxicity profile of irinotecan, e,g. myelosuppression and diarrhea. If a patient with UGT1A1*28 (7/7 homozygosity) is included in the low level of phase I period, the MTD of irinotecan might be set up in low dose without showing sufficient efficacy.

We think that it may be of deserve to evaluate the efficacy of paclitaxel and irinotecan combination regimen in gastric cancer patients and it is necessary to conduct phase I study to find out the accurate MTD of this regimen after considering the UGT1A1 polymorphism of patients.

So we designed this phase I/II study to evaluate the efficacy and toxicity of second-line chemotherapy with paclitaxel and irinotecan in fluoropyrimidine and platinum-pretreated advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* A patient who is able to walk and should have ECOG performance status of 0-1.
* Histologically confirmed adenocarcinoma of the stomach
* Unresectable locally advanced or initially metastatic or recurrent after curative resection
* Prior one regimen chemotherapy including fluoropyrimidine and platinum. (FP, XP, TS-1+cisplatin, FOLFOX)
* A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in Spiral CT or multidetector CT (MD CT), or 20 mm or longer in conventional CT (it should be used by a consistent method during the study period).
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it.
* A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* A patient with no measurable disease
* A patient with previous chemotherapy without containing fluoropyrimidine or platinum.
* A patient with UGT1A1*28 allele ((TA)7/7 homozygosity)
* A patient with previous active or passive immunotherapy.
* A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding
* A pregnant or lactating patient
* A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential.)
* A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study.
* A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of the skin and cervical carcinoma in situ are excluded.
* A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
* A patient with clinically significant (i.e. active) heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmias, etc) or myocardial infarction within past 12 months.
* A patient with interstitial pneumonia or diffused symptomatic fibrosis of the lungs.
* A patient with peripheral neuropathy of Grade 1 by NCI CTC, caused by other factors (e.g. alcohol, diabetes, etc). If the absence of deep tendon reflexes (DTRs) is the only neurologic disorder, this condition does not apply to the exclusion criteria.
* Organ allogenic transplantation requiring immunosuppressive therapy.
* A patient who developed uncontrolled serious infection or other uncontrolled serious concomitant diseases.
* A patient with moderate or severe renal insufficiency or serum creatinine > 1.5 X upper limit of normal].
* Adequate organ function
* A patient with hypersensitivity.
* A patient who has received major surgery within 4 weeks prior to the initiation of the study or a patient who is not completely recovered from impact of the major surgery.
* A patient who has participated in a clinical trial with other medications or therapy within 4 weeks prior to the initiation of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (phase I part) | during first cycle (first 3 week)
response rate (phase II part) | every 2 cycles response evaluation

SECONDARY OUTCOMES:
recommended phase II dose | after the determining MTD
time to progression | at the time of disease progression
overall survival | at the time of death
toxicities | every time of physical exam and laboratory evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea